CLINICAL TRIAL: NCT00533221
Title: Can Treatment With Human Growth Hormone Increase Strength in Spinal Muscular Atrophy Type II and III?
Brief Title: Pilot Study of Growth Hormon to Treat SMA Typ II and III
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Janbernd Kirschner, MD, University Hospital Freiburg
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMA-GH; 2005-002822-78
Record Dates: First submitted 2007-09-12; First posted 2007-09-21 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Muscular Atrophy, Spinal
Keywords: growth hormone; strength; Spinal muscular atrophy type II and III
MeSH Terms: conditions — Muscular Atrophy, Spinal; Spinal Muscular Atrophies of Childhood | interventions — Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Somatotropin (Active Comparator): subcutaneous application of somatotropin over 12 weeks followed by 8 weeks wash out period followed by 12 weeks subcutaneous placebo application
  Interventions: Drug: somatotropin
- Placebo (Placebo Comparator): 12 weeks placebo subcutaneous application followed by 8 weeks wash out and 12 weeks subcutaneous application of somatotropin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: somatotropin — 0,015 mg/kg/d as one dose s.c. in the evening over one week followed by a 11 week period with 0,03 mg/kg/d s.c. as one dose in the evening
  Other Names: Penfill®
  Arms: Somatotropin
Drug: Placebo — 0,015 mg/kg/d as one dose s.c. in the evening over one week followed by a 11 week period with 0,03 mg/kg/d s.c. as one dose in the evening
  Other Names: Penfill®
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Growth hormon can increase strength in spinal muscular atrophy type II and III.

DETAILED DESCRIPTION:
This pilot study is planned as a placebo-controlled cross-over trial in a limited number of patients. It is the aim to investigate the effect of GH on the short-term changes of strength and to investigate the tolerability of the treatment. If the results of the study are positive, further studies of longer duration addressing the development of motor function and quality of life could follow

ELIGIBILITY:
Inclusion Criteria:

* genetically confirmed diagnosis of Spinal Muscular Disease
* Spinal muscular atrophy type II or III
* age between 6 years and 35 years
* ability to perform the tests for measurement of muscle strength (handheld myometry)
* informed consent of the patient and/or parents

Exclusion Criteria:

* pregnancy or lactation
* woman with child bearing potential without contraception
* overweight or BMI over 30 kg/m²
* Treatment with other drugs, that can influence strength 8 weeks before participation in the study or during participation
* medical history or evidence of a malignant or cerebral tumor
* cardiovascular, intestinal, endocrinologically or airway disease
* Hypertension
* growth hormone deficiency
* hypersensitivity to one component part of the study medication
* participation on a clinical trial during the study or 3 month before
* abuse to drugs or alcohol
* patient incapable of contracting or not able to understand the character, meaning and consequences of the clinical trial

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2010-02 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Primary: sum of strength (hand held myometry) | 20 weeks

SECONDARY OUTCOMES:
Functional (time) tests, lung function, quality of life, | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Korinthenberg, Professor, Principal Investigator — University medical centre Freiburg, children's hospital
Locations (6):
- Germany (6):
  - von Haunersches Kinderspital, Munich, Bavaria
  - University Children'S Hospital, Göttingen, Lower Saxony
  - University Children'S Hospital, Essen, North Rhine-Westphalia
  - University Children'S Hospital, Mainz, Rhineland-Palatinate
  - University Children'S Hospital, Kiel, Schleswig-Holstein
  - Charité, Department of Neurpaediatrics, Berlin, State of Berlin

REFERENCES:
- [Result] Kirschner J, Schorling D, Hauschke D, Rensing-Zimmermann C, Wein U, Grieben U, Schottmann G, Schara U, Konrad K, Muller-Felber W, Thiele S, Wilichowski E, Hobbiebrunken E, Stettner GM, Korinthenberg R. Somatropin treatment of spinal muscular atrophy: a placebo-controlled, double-blind crossover pilot study. Neuromuscul Disord. 2014 Feb;24(2):134-42. doi: 10.1016/j.nmd.2013.10.011. Epub 2013 Nov 13. PMID 24300782
- See also: University Children's Hospital Freiburg, Germany — http://www.uniklinik-freiburg.de/kinderklinik